CLINICAL TRIAL: NCT00137735
Title: Gabapentin for Carpal Tunnel Syndrome: A Randomised Controlled Trial
Brief Title: Gabapentin for Carpal Tunnel Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IG-HK-GAB-01-02
Record Dates: First submitted 2005-08-29; First posted 2005-08-30 (Estimated); Last update posted 2007-10-31 (Estimated); Status verified 2007-10

CONDITIONS: Carpal Tunnel Syndrome
Keywords: carpal tunnel syndrome; gabapentin
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Active Comparator): Gabapentin
  Interventions: Drug: Gabapentin
- 2 (Placebo Comparator): Placebo
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Gabapentin — 300mg tds
  Arms: 1
Other: placebo — tds
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether gabapentin is safe and effective in the treatment of carpal tunnel syndrome (CTS).

DETAILED DESCRIPTION:
A variety of treatment options exist at present for carpal tunnel syndrome (CTS) with no universal agreement. Recent reports suggested that untreated CTS might improve or remain stationary. In this respect, treatment directing towards symptom suppression alone may have a role in the initial management of CTS. Gabapentin (1-[aminomethyl]-cyclohexaneacetic acid; Neurontin, Pfizer) is an effective drug for treatment of neuropathic pain and has been reported to be effective in case series for the treatment of CTS with relatively benign side effects profile. The purpose of this study was to evaluate the safety and efficacy of gabapentin in the treatment of CTS.

ELIGIBILITY:
Inclusion Criteria:

* Sensory symptoms over median nerve distribution for more than three months.
* Confirmatory electrophysiologic results defined as prolonged median nerve distal motor latencies (DML) > 4 ms or median-ulnar palmer sensory latency differences > 0.5 ms.

Exclusion Criteria:

* Patients with evidence of severe CTS: fibrillation potentials or reinnervation on needle examination of the abductor pollicis brevis muscle or clinical examination showing wastage of the thenar muscles. (These patients were referred for surgical decompression on presentation.)
* Clinical or electrophysiological evidence of accompanying conditions that could mimic CTS or interfere with its evaluation, such as proximal median neuropathy, cervical radiculopathy, or significant polyneuropathy.
* Known epilepsy.
* Patients who have received previous steroid injection or oral steroid therapy for CTS.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2003-10; Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Global symptom score (GSS) recorded by a physician blinded to the allocation of treatment at 8 weeks | 8 weeks

SECONDARY OUTCOMES:
GSS at 2 weeks | 2 weeks
Grip strength as functional assessment at 2 and 8 weeks | 2 weeks, 8 weeks
Tolerability | throughout subject's participation in trial

CONTACTS AND LOCATIONS:
Overall Officials: Andrew CF Hui, FHKAM, Principal Investigator — Department of Medicine & Therapeutics, Faculty of Medicine, The Chinese University of Hong Kong
Locations (2):
- Hong Kong (2):
  - Prince of Wales Hospital, Shatin, New Territories
  - North District Hospital, Sheung Shui, New Territories